CLINICAL TRIAL: NCT00697749
Title: Phase III Study to Compare Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Novel Adjuvanted Hepatitis B Vaccine Adminstered Intramuscularly, According to a 0, 6 Month Schedule, to Engerix™-B 20 mcg Administered According to a 0,1,6 Month Schedule in Healthy Volunteers Positive for the HLA-DQ2 Genotype
Brief Title: Immunogenicity and Safety of a Novel Adjuvanted HBV Vaccine in Healthy Volunteers Positive for the HLA-DQ2 Genotype
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208129/034
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Recombinant hepatitis B vaccine; Adjuvanted hepatitis B vaccine; Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 2-dose intramuscular injection
  Arms: Group A
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group B

SUMMARY:
This study compares the immunogenicity and safety of the novel adjuvanted HBV vaccine and Engerix™-B administered to subjects who were positively identified as having the HLA-DQ2 genotype

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* A male or female ≥ 15 years of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the subject/ from the parents or guardians of the subject.
* Known to be seronegative for anti-HBs-antibodies, anti-HBc-antibodies and/or HBsAg.
* Positive for the HLA-DQ2 genotype as determined in the previous sero-HBV-069 prevalence study.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or use adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Previous vaccination against hepatitis B.
* History of non-response to previous hepatitis B vaccination.
* Known exposure to hepatitis B within 6 weeks.
* History of hepatitis B infection.
* Confirmed human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration/ administration during the study period.
* Pregnant or lactating female

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 1999-04; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At month 7

SECONDARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general signs and symptoms | During a 4 day follow-up period after each vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | During a 30 day follow-up period after each vaccination
Occurrence, intensity and relationship to vaccination of serious adverse events (SAEs) | During the study period
Anti-HBs antibody concentrations | Day 0, Month 1, Month 6 and Month 7
Cell mediated immunity | At Months 0 and 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208129/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register